CLINICAL TRIAL: NCT02189473
Title: Radiotherapy of Motor Deficits From Metastatic Epidural Spinal Cord Compression (10 x 3 Gy Versus 5 x 4 Gy)
Brief Title: Radiotherapy of Motor Deficits From Metastatic Epidural Spinal Cord Compression
Acronym: SCORE-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dirk Rades, MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Dirk Rades, MD, Prof. Dr. Dirk Rades. MD, University Hospital Schleswig-Holstein
Organization: University Hospital Schleswig-Holstein (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARO 200901
Record Dates: First submitted 2014-07-07; First posted 2014-07-14 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-02

CONDITIONS: Metastatic Epidural Spinal Cord Compression
Keywords: metastatic epidural spinal cord compression; motor function; ambulatory status; pain; quality of life; overall survival; local control; toxicity
MeSH Terms: conditions — Pain | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5 x 4 Gy in 1 week (Experimental): radiotherapy with 5 x 4 Gy in 1 week (5 x 4 Gy per week)
  Interventions: Radiation: radiotherapy
- 10 x 3 Gy in 2 weeks (Active Comparator): radiotherapy with 10 x 3 Gy in 2 weeks (5 x 3 Gy per week)
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — external beam radiotherapy (5 x 4 Gy versus 10 x 3 Gy)

SUMMARY:
The primary aim of this randomized multi-center trial is to investigate the efficacy of the radiotherapy regimens 5 x 4 Gy and 10 x 3 Gy with respect to the effect on motor function in patients with metastatic epidural spinal cord compression.

DETAILED DESCRIPTION:
The primary aim of this randomized multi-center trial is to investigate the efficacy of the radiotherapy regimens 5 x 4 Gy and 10 x 3 Gy with respect to the effect on motor function in patients with metastatic epidural spinal cord compression. The response rate (improvement in motor function or prevention of progression) will be assessed at one month following radiotherapy.

In addition, the following endpoints will be evaluated:

1. Motor function; additional assessments directly and at 3 and at 6 months after radiotherapy
2. Ability to walk; assessment directly and at 1, 3 and 6 months after radiotherapy
3. Sensory function; assessment directly and at 1, 3 and 6 months after radiotherapy
4. Quality of life; evaluation directly and at 1, 3 and 6 months after radiotherapy
5. Pain assessment directly and at 1, 3 and 6 months after radiotherapy
6. Overall survival up to 6 months following radiotherapy
7. Local Progression-free survival up to 6 months following radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Motor deficits of the lower extremities resulting from metastatic epidural spinal cord compression, which have persisted for no longer than 30 days
* Confirmation of diagnosis by magnetic resonance imaging (spinal computed tomography allowed)
* Relatively poor survival prognosis (defined as ≤35 points on the survival score published in Cancer 2008)
* Written informed consent

Exclusion Criteria:

* Prior radiotherapy or surgery of the spinal areas affected by MESCC
* History of symptomatic brain tumor or symptomatic brain metastases
* Metastases of the cervical spine only
* Other severe neurological disorders
* Pregnancy, Lactation
* Indication for decompressive surgery + stabilization of the affected spinal areas

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2010-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Rades, MD, Study Chair — Department of Radiation Oncology, University of Lübeck, Germany
Locations (15):
- Mayo Clinic, Scottsdale, Arizona, United States
- Germany (9):
  - Oberschwabenklinik Ravensburg, Ravensburg, Baden-Wutemberg
  - Klinikum Bayreuth, Bayreuth, Bavaria
  - University of Regensburg, Regensburg, Bavaria
  - University of Würzburg, Würzburg, Bavaria
  - Ruhr University, Bochum, North Rhine-Westphalia
  - Radiotherapy Practice Dresden-Friedrichstadt, Dresden, Saxony
  - University of Lübeck, Lübeck, Schleswig-Holstein
  - Charite Berlin, Berlin
  - Center of Radiotherapy and Radiation Oncology, Bremen
- Institute of Oncology, Vilnius University, Vilnius, Lithuania
- Saad Specialist Hospital, Khobar, Saudi Arabia
- Institute of Oncology, Ljubljana, Slovenia
- Spain (2):
  - Consorcio Hospitalario Provencial de Castellon, Valencia, Castellon
  - Cruces University Hospital, Barakaldo, Vizcaya (Basque Country)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maranzano E, Latini P. Effectiveness of radiation therapy without surgery in metastatic spinal cord compression: final results from a prospective trial. Int J Radiat Oncol Biol Phys. 1995 Jul 15;32(4):959-67. doi: 10.1016/0360-3016(95)00572-g. PMID 7607970
- [Background] Sorensen S, Borgesen SE, Rohde K, Rasmusson B, Bach F, Boge-Rasmussen T, Stjernholm P, Larsen BH, Agerlin N, Gjerris F, et al. Metastatic epidural spinal cord compression. Results of treatment and survival. Cancer. 1990 Apr 1;65(7):1502-8. doi: 10.1002/1097-0142(19900401)65:73.0.co;2-d. PMID 2311062
- [Background] Helweg-Larsen S, Sorensen PS, Kreiner S. Prognostic factors in metastatic spinal cord compression: a prospective study using multivariate analysis of variables influencing survival and gait function in 153 patients. Int J Radiat Oncol Biol Phys. 2000 Mar 15;46(5):1163-9. doi: 10.1016/s0360-3016(99)00333-8. PMID 10725627
- [Background] Leviov M, Dale J, Stein M, Ben-Shahar M, Ben-Arush M, Milstein D, Goldsher D, Kuten A. The management of metastatic spinal cord compression: a radiotherapeutic success ceiling. Int J Radiat Oncol Biol Phys. 1993 Sep 30;27(2):231-4. doi: 10.1016/0360-3016(93)90232-k. PMID 8407396
- [Background] Rades D, Blach M, Bremer M, Wildfang I, Karstens JH, Heidenreich F. Prognostic significance of the time of developing motor deficits before radiation therapy in metastatic spinal cord compression: one-year results of a prospective trial. Int J Radiat Oncol Biol Phys. 2000 Dec 1;48(5):1403-8. doi: 10.1016/s0360-3016(00)01408-5. PMID 11121640
- [Background] Rades D, Heidenreich F, Bremer M, Karstens JH. Time of developing motor deficits before radiotherapy as a new and relevant prognostic factor in metastatic spinal cord compression: final results of a retrospective analysis. Eur Neurol. 2001;45(4):266-9. doi: 10.1159/000052141. PMID 11385267
- [Background] Rades D, Heidenreich F, Karstens JH. Final results of a prospective study of the prognostic value of the time to develop motor deficits before irradiation in metastatic spinal cord compression. Int J Radiat Oncol Biol Phys. 2002 Jul 15;53(4):975-9. doi: 10.1016/s0360-3016(02)02819-5. PMID 12095565
- [Background] Arcangeli G, Giovinazzo G, Saracino B, D'Angelo L, Giannarelli D, Arcangeli G, Micheli A. Radiation therapy in the management of symptomatic bone metastases: the effect of total dose and histology on pain relief and response duration. Int J Radiat Oncol Biol Phys. 1998 Dec 1;42(5):1119-26. doi: 10.1016/s0360-3016(98)00264-8. PMID 9869238
- [Background] Niewald M, Tkocz HJ, Abel U, Scheib T, Walter K, Nieder C, Schnabel K, Berberich W, Kubale R, Fuchs M. Rapid course radiation therapy vs. more standard treatment: a randomized trial for bone metastases. Int J Radiat Oncol Biol Phys. 1996 Dec 1;36(5):1085-9. doi: 10.1016/s0360-3016(96)00388-4. PMID 8985030
- [Background] 8 Gy single fraction radiotherapy for the treatment of metastatic skeletal pain: randomised comparison with a multifraction schedule over 12 months of patient follow-up. Bone Pain Trial Working Party. Radiother Oncol. 1999 Aug;52(2):111-21. PMID 10577696
- [Background] Steenland E, Leer JW, van Houwelingen H, Post WJ, van den Hout WB, Kievit J, de Haes H, Martijn H, Oei B, Vonk E, van der Steen-Banasik E, Wiggenraad RG, Hoogenhout J, Warlam-Rodenhuis C, van Tienhoven G, Wanders R, Pomp J, van Reijn M, van Mierlo I, Rutten E. The effect of a single fraction compared to multiple fractions on painful bone metastases: a global analysis of the Dutch Bone Metastasis Study. Radiother Oncol. 1999 Aug;52(2):101-9. doi: 10.1016/s0167-8140(99)00110-3. PMID 10577695
- [Background] Rades D, Stalpers LJ, Veninga T, Schulte R, Hoskin PJ, Obralic N, Bajrovic A, Rudat V, Schwarz R, Hulshof MC, Poortmans P, Schild SE. Evaluation of five radiation schedules and prognostic factors for metastatic spinal cord compression. J Clin Oncol. 2005 May 20;23(15):3366-75. doi: 10.1200/JCO.2005.04.754. PMID 15908648
- [Background] Emami B, Lyman J, Brown A, Coia L, Goitein M, Munzenrider JE, Shank B, Solin LJ, Wesson M. Tolerance of normal tissue to therapeutic irradiation. Int J Radiat Oncol Biol Phys. 1991 May 15;21(1):109-22. doi: 10.1016/0360-3016(91)90171-y. PMID 2032882
- [Background] Barendsen GW. Dose fractionation, dose rate and iso-effect relationships for normal tissue responses. Int J Radiat Oncol Biol Phys. 1982 Nov;8(11):1981-97. doi: 10.1016/0360-3016(82)90459-x. No abstract available. PMID 6759484
- [Background] Koswig S, Budach V. [Remineralization and pain relief in bone metastases after after different radiotherapy fractions (10 times 3 Gy vs. 1 time 8 Gy). A prospective study]. Strahlenther Onkol. 1999 Oct;175(10):500-8. doi: 10.1007/s000660050061. German. PMID 10554645
- [Background] Rades D, Dunst J, Schild SE. The first score predicting overall survival in patients with metastatic spinal cord compression. Cancer. 2008 Jan 1;112(1):157-61. doi: 10.1002/cncr.23150. PMID 17948910
- [Background] Tomita T, Galicich JH, Sundaresan N. Radiation therapy for spinal epidural metastases with complete block. Acta Radiol Oncol. 1983;22(2):135-43. doi: 10.3109/02841868309134353. PMID 6310968
- [Background] Maranzano E, Bellavita R, Rossi R, De Angelis V, Frattegiani A, Bagnoli R, Mignogna M, Beneventi S, Lupattelli M, Ponticelli P, Biti GP, Latini P. Short-course versus split-course radiotherapy in metastatic spinal cord compression: results of a phase III, randomized, multicenter trial. J Clin Oncol. 2005 May 20;23(15):3358-65. doi: 10.1200/JCO.2005.08.193. Epub 2005 Feb 28. PMID 15738534
- [Derived] Rades D, Segedin B, Conde-Moreno AJ, Ferrer-Albiach C, Metz M, Polat B, Badakhshi H, Schreiber A, Nitsche M, Cacicedo J, Schild SE. Patient-Reported Outcomes-Secondary Analysis of the SCORE-2 Trial Comparing 4 Gy x 5 to 3 Gy x 10 for Metastatic Epidural Spinal Cord Compression. Int J Radiat Oncol Biol Phys. 2019 Nov 15;105(4):760-764. doi: 10.1016/j.ijrobp.2019.08.002. Epub 2019 Aug 12. PMID 31415797
- [Derived] Rades D, Segedin B, Conde-Moreno AJ, Garcia R, Perpar A, Metz M, Badakhshi H, Schreiber A, Nitsche M, Hipp P, Schulze W, Adamietz IA, Norkus D, Rudat V, Cacicedo J, Schild SE. Radiotherapy With 4 Gy x 5 Versus 3 Gy x 10 for Metastatic Epidural Spinal Cord Compression: Final Results of the SCORE-2 Trial (ARO 2009/01). J Clin Oncol. 2016 Feb 20;34(6):597-602. doi: 10.1200/JCO.2015.64.0862. Epub 2016 Jan 4. PMID 26729431

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5 x 4 Gy in 1 Week | 10 x 3 Gy in 2 Weeks
Started | 101 | 102
Completed | 78 | 77
Not Completed | 23 | 25
Not completed — Death | 22 | 23
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 x 4 Gy in 1 Week | 10 x 3 Gy in 2 Weeks | Total
Number analyzed (Participants) | 101 | 102 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 39 | 34 | 73
  >=65 years | 62 | 67 | 129
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 38 | 79
  Male | 60 | 64 | 124
Region of Enrollment [Number; unit: participants]
  Slovenia | 8 | 9 | 17
  Lithuania | 1 | 0 | 1
  Germany | 75 | 89 | 164
  Spain | 17 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Showing Improvement or no Further Progression of Motor Deficits at 1 Month Following Radiotherapy
Description: Overall response was defined as improvement or no further progression of motor deficits following radiotherapy.
  Motor function was graded with the following 8-point scale: 0, complete paraplegia; 1, palpable or visible muscle contractions; 2, active movement of the leg without gravity; 3, active movement against gravity; 4, active movement against mild resistance; 5, active movement against intermediate resistance; 6, active movement against strong resistance; and 7, normal strength.
  Motor function was recorded separately for each leg resulting in total points of 0 to 14. Improvement of motor function was defined as an increase by at least 2 points compared to baseline. No further progression was defined as +/-1 point (i.e. +1 point, +/- 0 points or -1 point).
Time Frame: at 1 month following radiotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | 5 x 4 Gy in 1 Week | 10 x 3 Gy in 2 Weeks
Number analyzed (Participants) | 78 | 77
Participants | 68 | 69

2. Secondary Outcome: Number of Participants Who Were Able to Walk at 1 Month Following Radiotherapy
Description: Ambulatory status was assessed using the following scoring system:
  0 = Normal strength
  1. = Ambulatory without aid
  2. = Ambulatory with aid
  3. = Not ambulatory
  A patient with a score equal to or less than 2 is considered "able to walk". Both participants that could and could not walk prior to radiotherapy have been included in this assessment..
Time Frame: at 1 month following radiotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | 5 x 4 Gy in 1 Week | 10 x 3 Gy in 2 Weeks
Number analyzed (Participants) | 78 | 77
Participants | 56 | 57

3. Secondary Outcome: Number of Participants Who Were Alive at 6 Months Following Radiotherapy Without Deterioration of Motor Function During (or Directly Following) Radiotherapy and Freedom From In-field Recurrence of Metastatic Spinal Cord Compression Following Radiotherapy
Description: Local Progression Free Survival (LPFS) was defined as freedom from progression of motor deficits during or one month following radiotherapy and freedom from in-field recurrence of metastatic spinal cord compression (MSCC) following radiotherapy.
  An in-field recurrence was defined as a recurrence of MSCC associated with motor deficits in the region of the spinal cord that had been previously irradiated for MSCC.
  In case of clinical suspicion of sich a recurrence, a spinal MRI was performed to confirm the diagnosis. Time to in-field recurrence was calculated from the last day of radiotherapy, and the patients were followed for a maximum of 6 months after the end of radiotherapy. The values of 6-month LPFS were estimated using the Kaplan-Meier method.
Time Frame: 6 months following radiotherapy
Measure: Number; unit: Percentage of participants
Arm/Group | 5 x 4 Gy in 1 Week | 10 x 3 Gy in 2 Weeks
Number analyzed (Participants) | 101 | 102
Percentage of participants | 75.2 | 81.8

4. Secondary Outcome: Number of Participants Who Experienced Relief of Distress at 1 Month Following Radiotherapy Compared to Baseline
Description: Distress (as an indicator of impairment of quality of life) was measured with the distress-thermometer. the patients rated their level of distress on a scale ranging from 0 (no distress) to 10 (extreme distress). Patients rated the distress they experienced during the last week and stated the reasons for distress from a list of items.
  An improvement (lower score) by 2 points was considered a clinically relevant relief of distress. Patients with baseline-scores of 0-1 points were not included, since improvement by 2 points was not possible.
Time Frame: at 1 month following radiotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | 5 x 4 Gy in 1 Week | 10 x 3 Gy in 2 Weeks
Number analyzed (Participants) | 74 | 75
Participants | 43 | 47

5. Secondary Outcome: Number of Participants Who Experienced Relief of Pain at 1 Month Following Radiotherapy Compared to Baseline
Description: Pain was measured with a numeric self-rating scale ranging from 0 (no pain) to 10 (worst pain).
  Relief of pain was defined as improvement (=decrease of pain) by at least 2 points without increase of analgesics. Patients with baseline-scores of 0-1 points were not included, since improvement by 2 points was not possible.
Time Frame: at 1 month following radiotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | 5 x 4 Gy in 1 Week | 10 x 3 Gy in 2 Weeks
Number analyzed (Participants) | 68 | 70
Participants | 36 | 40

6. Secondary Outcome: Number of Participants Who Were Alive at 6 Months Following Radiotherapy
Description: Overall Survival (OS) was defined as freedom from death of any cause.
  Time to death was calculated from the last day of radiotherapy, and the patients were followed for a maximum of 6 months after the end of radiotherapy. The values of 6-month OS were estimated using the Kaplan-Meier method.
Time Frame: 6 months following radiotherapy
Measure: Number; unit: Percentage of participants
Arm/Group | 5 x 4 Gy in 1 Week | 10 x 3 Gy in 2 Weeks
Number analyzed (Participants) | 101 | 102
Percentage of participants | 42.3 | 37.8

7. Secondary Outcome: Number of Participants Showing Improvement of Motor Deficits at 1 Month Following Radiotherapy
Description: Motor function was graded with the following 8-point scale: 0, complete paraplegia; 1, palpable or visible muscle contractions; 2, active movement of the leg without gravity; 3, active movement against gravity; 4, active movement against mild resistance; 5, active movement against intermediate resistance; 6, active movement against strong resistance; and 7, normal strength.
  Motor function was recorded separately for each leg resulting in total points of 0 to 14. Improvement of motor function was defined as an increase by at least 2 points compared to baseline.
Time Frame: at 1 month following radiotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | 5 x 4 Gy in 1 Week | 10 x 3 Gy in 2 Weeks
Number analyzed (Participants) | 78 | 77
Participants | 30 | 34

8. Secondary Outcome: Number of Participants Experiencing at Least One Grade >=2 Radiotherapy-related Toxicity
Description: Toxicity was assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) (version 4)
Time Frame: during radiotherapy and up to 6 months following radiotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | 5 x 4 Gy in 1 Week | 10 x 3 Gy in 2 Weeks
Number analyzed (Participants) | 101 | 102
Participants
  at least 1 grade >=2 radiotherapy-related toxicity | 11 | 15
  no grade >=2 radiotherapy-related toxicity | 90 | 87

ADVERSE EVENTS:
Arm/Group | 5 x 4 Gy in 1 Week | 10 x 3 Gy in 2 Weeks
All-Cause Mortality (participants affected / at risk) | 58/101 | 62/102
Serious Adverse Events (participants affected / at risk) | 12/101 | 7/102
Other Adverse Events (participants affected / at risk) | 25/101 | 26/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 x 4 Gy in 1 Week (N=101) | 10 x 3 Gy in 2 Weeks (N=102)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
sepsis (Infections and infestations) | 2 (2) | 2 (2)
pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0)
subdural bleeding (Nervous system disorders) | 1 (1) | 0 (0)
acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
reflux esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
desorientation (Nervous system disorders) | 1 (1) | 0 (0)
infection (Infections and infestations) | 0 (0) | 2 (2)
gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thrombopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
hypotonia (General disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 x 4 Gy in 1 Week (N=101) | 10 x 3 Gy in 2 Weeks (N=102)
nausea/vomiting (Gastrointestinal disorders) | 16 (21) | 20 (21)
diarrhea (Gastrointestinal disorders) | 5 (8) | 8 (8)
fatigue (General disorders) | 3 (4) | 5 (6)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
radiation dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
constipation (Gastrointestinal disorders) | 1 (1) | 1 (2)
gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
cachexia (General disorders) | 1 (2) | 0 (0)
increased levels of transaminases (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes